CLINICAL TRIAL: NCT07058259
Title: The Effect of Acupuncture in COPD Patients With Persistent Dyspnea Despite Medical Treatment
Brief Title: Acupuncture for Persistent Dyspnea Despite Medical Treatment in COPD
Acronym: COPD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Bilinç Doğruöz Karatekin, MD, Specialist of PMR,Principal Investigator, Istanbul Medeniyet University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MU Acupuncture and COPD
Record Dates: First submitted 2025-06-22; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-06

CONDITIONS: COPD (Chronic Obstructive Pulmonary Disease); Acupuncture
Keywords: COPD; ACUPUNCTURE; dyspnea; chronic obstructive pulmonary disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea | interventions — Acupuncture Therapy; laminin A

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard COPD Pharmacological Treatment Group (Control) (Active Comparator): Drug: Standard COPD Pharmacological Therapy (LAMA + LABA or LAMA + LABA + ICS) Patients receive standard pharmacological treatment for COPD according to current clinical guidelines without acupuncture. This will serve as a control group.
  Interventions: Drug: Standard COPD Pharmacological Therapy (LAMA + LABA or LAMA + LABA + ICS)
- Acupuncture + Standard COPD Pharmacological Treatment Group (Intervention) (Experimental): Participants in this group will receive standard pharmacological treatment for COPD in addition to acupuncture therapy. - Standard COPD Pharmacological Therapy (LAMA + LABA or LAMA + LABA + ICS)
  Acupuncture will be administered twice weekly for 5 weeks (10 sessions total) at predefined bilateral acupoints: LU1, LU9, LI18, ST36, GB12, BL13, BL20, and BL23. Single-use, sterile 25 mm × 0.25 mm needles will be inserted at each point for 20 minutes per session.
  Interventions: Behavioral: Acupuncture; Drug: Standard COPD Pharmacological Therapy (LAMA + LABA or LAMA + LABA + ICS)

INTERVENTIONS:
Behavioral: Acupuncture — Acupuncture will be administered twice weekly for 5 weeks (10 sessions total) at predefined bilateral acupoints: LU1, LU9, LI18, ST36, GB12, BL13, BL20, and BL23. Single-use, sterile 25 mm × 0.25 mm needles will be inserted at each point for 20 minutes per session.
  Arms: Acupuncture + Standard COPD Pharmacological Treatment Group (Intervention)
Drug: Standard COPD Pharmacological Therapy (LAMA + LABA or LAMA + LABA + ICS) — Patients in this group receive standard pharmacological treatment for COPD according to current clinical guidelines. Treatment includes either dual or triple inhaler therapy:
  Dual Therapy (LABA + LAMA): Patients receive a long-acting beta-agonist (LABA) such as Formoterol, Salmeterol, Olodaterol, Vilanterol, or Indacaterol, in combination with a long-acting muscarinic antagonist (LAMA) such as Tiotropium bromide, Umeclidinium, or Glycopyrronium.
  Triple Therapy (LABA + LAMA + ICS): Patients receive the above combination of LABA and LAMA plus an inhaled corticosteroid (ICS) such as Budesonide, Fluticasone, or Beclometasone.
  These medications may be administered either as fixed-dose combination inhalers or as separate inhalers, depending on patient needs and physician discretion. The treatment regimen is individualized based on clinical condition, prior therapy, and symptom severity.
  Other Names: Dual therapy (LAMA+LABA); Triple Therapy (LAMA+LABA+ICS)

SUMMARY:
This randomized controlled trial aims to evaluate the effectiveness of acupuncture as an adjunctive non-pharmacological therapy in patients with stable COPD who continue to experience dyspnea despite optimal medical treatment.

DETAILED DESCRIPTION:
A total of 60 patients diagnosed with COPD will be randomly assigned to either a control group receiving standard pharmacological treatment or an intervention group receiving standard treatment plus acupuncture. The intervention group will undergo 10 acupuncture sessions (twice weekly for 5 weeks) using predefined acupuncture points based on previous COPD studies.

Primary outcomes include changes in dyspnea severity measured by the Modified Medical Research Council (mMRC) Dyspnea Scale, the COPD Assessment Test (CAT), and the Borg scale. Secondary outcomes include changes in pulmonary function (FEV1, FVC, FEV1/FVC) and functional exercise capacity assessed by the 6-Minute Walk Test (6MWT) and Incremental Shuttle Walk Test (ISWT). Spirometry and exercise testing will be performed pre- and post-intervention. The study will help determine whether acupuncture provides statistically and clinically meaningful improvements in symptom burden and exercise tolerance in COPD management.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers aged between 40 and 80 years, who are communicative and cooperative,
* Diagnosed with COPD for at least 3 months,
* Receiving dual or triple regular pharmacological therapy for at least 3 months,
* Post-bronchodilator FEV1/FVC <70% and predicted FEV1 <80% on spirometry, mMRC (Modified Medical Research Council) dyspnea score of 2 or higher,
* COPD Assessment Test (CAT) score of 10 or higher.

Exclusion Criteria:

* Patients who do not consent to participate in the study,
* Patients with communication difficulties or with visual, walking, or hearing impairments,
* Patients currently experiencing a COPD exacerbation or with a history of exacerbation within the past month,
* Patients with Stage 1 COPD (FEV1 ≥ 80%),
* COPD patients receiving monotherapy,
* Patients with mMRC score <2 and CAT score <10,
* Patients with unstable angina, acute myocardial infarction (within 3-5 days), uncontrolled arrhythmia, active endocarditis, acute myocarditis/pericarditis, symptomatic severe aortic stenosis, lower extremity DVT, uncontrolled asthma/COPD, pulmonary edema, oxygen saturation (SpO₂) ≤ 90%, acute respiratory failure, or suspected dissecting aneurysm,
* Patients receiving long-term oxygen therapy (LTOT),
* COPD patients who have experienced more than two exacerbations in the past year.

Withdrawal Criteria:

* Patients who are unable to complete acupuncture sessions or follow-up assessments in the control group for any reason,
* Patients who experience an exacerbation during the study (they will be reassessed one month after recovery and may be re-included if eligible),
* Patients who miss more than two acupuncture sessions.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Modified Medical Research Council (mMRC) Dyspnea Scale | From baseline to the end of treatment at 6 weeks
  Change in dyspnea severity measured by the Modified Medical Research Council (mMRC) Dyspnea Scale from baseline to 6 weeks.

SECONDARY OUTCOMES:
COPD Assessment Test (CAT) | From baseline to the end of treatment at 6 weeks
  Change in COPD Assessment Test (CAT) score.The CAT score evaluates overall symptom burden and quality of life in COPD patients.
Change in Forced Expiratory Volume in 1 Second (FEV1) | From baseline to the end of treatment at 6 weeks
  FEV1 will be measured via spirometry pre- and post-bronchodilator to assess lung function
6-Minute Walk Test (6MWT) | From baseline to the end of treatment at 6 weeks
  Change in exercise capacity measured by the 6-Minute Walk Test (6MWT) distance
Incremental Shuttle Walk Test (ISWT) | From baseline to the end of treatment at 6 weeks
  Change in exercise tolerance assessed by the Incremental Shuttle Walk Test (ISWT)
Change in Forced Vital Capacity (FVC) | From baseline to the end of treatment at 6 weeks
  FVC will be measured via spirometry pre- and post-bronchodilator to assess pulmonary capacity.
Change in FEV1/FVC Ratio | From baseline to the end of treatment at 6 weeks
  The FEV1/FVC ratio will be calculated from spirometry values to evaluate airway obstruction severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medeniyet University Faculty of Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No